CLINICAL TRIAL: NCT01793064
Title: An Adaptive Physical Activity Intervention for Overweight Adults: A Randomized Controlled Trial
Brief Title: An Adaptive Physical Activity Intervention for Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Active Living Research (Other)
Responsible Party: Principal Investigator, Marc Adams, Assistant Professor, Exercise and Wellness Program, School of Nutrition and Health Promotion, College of Health Solutions., Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AD-31475
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Physical Activity
Keywords: Pedometer,; adaptive,; exercise,; reinforcement,; goal setting,; technology,; email,; weight loss; mHealth; eHealth
MeSH Terms: conditions — Motor Activity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adaptive Intervention Group (AI) (Experimental): Adaptive Intervention Group (AI) receives adaptive step goals and feedback/incentives based on personal physical activity performance.
  Interventions: Behavioral: Adaptive Intervention (AI)
- Static Intervention group (SI) (Active Comparator): Static Intervention group (SI) receives a static "usual care" goal of 10,000 steps/day and feedback/incentives for uploading their pedometer to the study website.
  Interventions: Behavioral: Static Intervention (SI)

INTERVENTIONS:
Behavioral: Adaptive Intervention (AI) — Adaptive Intervention Group (AI) receives adaptive step goals and feedback/incentives based on personal physical activity performance.
  Arms: Adaptive Intervention Group (AI)
Behavioral: Static Intervention (SI) — Static Intervention group (SI) receives a static "usual care" goal of 10,000 steps/day and feedback/incentives for uploading their pedometer to the study website.
  Arms: Static Intervention group (SI)

SUMMARY:
The purpose of this study is to develop and evaluate an adaptive shaping intervention based on Behavioral Economics and Operant principles to promote physical activity behaviors (adaptive group) and compare to a static physical activity intervention (static group) using a two-group randomized controlled trial design. Participants will include 20 overweight men and women (BMI 25-35 kg/m2) between 18 to 55 years. Both groups will receive the following components: 1) a pedometer, 2) self-monitoring of physical activity, 3) brief educational materials, 4) motivational prompts, 5) physical activity goals, and 6) small financial incentives. The Adaptive Intervention (AI) group will receive adaptive goals and feedback based on percentiles and a "moving" window of their recent physical activity, with incentives linked to goal attainment. Comparison intervention participants will receive the static 10,000 steps per day goal, with matching incentive amounts but without incentives linked to goal attainment. The study will compare differences in goal setting and shaping procedures that aim to increase physical activity behavior.

Primary aims include:

1. To determine whether physical activity (pedometer-measured steps/day) in both the Adaptive and Static interventions increased compared to their respective baselines. Hypothesis: Both the adaptive and static interventions will result in increased physical activity over 6 months.
2. To evaluate whether the Adaptive Intervention results in greater change in physical activity (pedometer-measured steps/day) compared to the Static Intervention. Hypothesis: The adaptive intervention will result in significantly greater physical activity, measured by pedometer, compared to the static intervention over 6 months.
3. To assess participants' satisfaction with the overall program. Hypothesis: Adaptive Intervention participants will report greater overall satisfaction with the intervention than the Static Intervention participants.

ELIGIBILITY:
Inclusion Criteria:

1. Live in San Diego County.
2. Be between 18 and 55 years old.
3. Currently not exceeding 1,000 MET-minutes per week of physical activity determined by the International Physical Activity Questionnaire (IPAQ short form).
4. Not suffering from a medical condition or taking medication(s) that would prohibit one from adopting a moderate intensity physical activity program.
5. Have a body mass index between 25 and 35 kg/m2.
6. Not currently pregnant.
7. Familiar with email and access to email and the internet daily,
8. Not planning to leave San Diego County for more than 10 days over the next 6 months.
9. Not planning to move away from San Diego County in the next 6 months.
10. Potential participants must have access to Microsoft Windows (XP, Vista, or windows 7) on a daily basis. If they do not, they would need to have daily access to and use Windows virtualization software (e.g. Parallels, VMware) for an Apple operating system.

Exclusion Criteria:

1. Does not live in Dan Diego.
2. Individuals under the age of 18 or over 55.
3. Those who exceed 1,000 met-minutes of physical activity per week determined by the International Physical Activity Questionnaire (IPAQ short form).
4. Suffering from a medical condition or taking medication which will prohibit one from adopting a moderate intensity physical activity program.
5. Does not have a BMI between 25 and 35 kg/m2.
6. Currently Pregnant.
7. Unfamiliar with email, or does not have access to the internet and email daily.
8. Planning to leave San Diego for more than ten days.
9. Planning to move from San Diego in the next 6 months.
10. Does not have access to Microsoft Windows or a Windows virtualization software for an Apple operating system.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Physical activity measured daily over 6 months by Omron pedometers (HJ-720ITC) . | 6 months
  Participants in both groups will be provided an Omron (HJ-720ITC) pedometer on the first day of the baseline phase, and will continue to use the pedometer throughout the entire study.

SECONDARY OUTCOMES:
Satisfaction Survey | 6 months
  At the end of the intervention phase, participants completed a satisfaction interview to rate on Likert-type scales and open-ended questions how motivating or burdensome specific study components were to them, their overall satisfaction with the study, personal experience with the intervention, any side effects or injuries, and their recommendations for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Adams, PhD, Principal Investigator — Arizona State University
Locations (1):
- San Diego State University, San Diego, California, United States

REFERENCES:
- [Result] Adams MA, Sallis JF, Norman GJ, Hovell MF, Hekler EB, Perata E. An adaptive physical activity intervention for overweight adults: a randomized controlled trial. PLoS One. 2013 Dec 9;8(12):e82901. doi: 10.1371/journal.pone.0082901. eCollection 2013. PMID 24349392